CLINICAL TRIAL: NCT01836042
Title: Post-approval Study of The Glaukos® iStent® Trabecular Micro-bypass Stent System In Conjunction With Cataract Surgery: Extended Follow-up of the Premarket Cohort
Brief Title: Post-approval Study of The Glaukos® iStent® Trabecular Micro-bypass Stent: Extended Follow-up of the Premarket Cohort
Status: Completed | Type: Observational
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: GTS100-PAS
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary open-angle glaucoma (POAG); Trabecular meshwork; iStent
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Randomized iStent: Implantation of one iStent in conjunction with cataract surgery, patients randomized to group
- Randomized cataract surgery: Cataract surgery alone, patients randomized to group
- Non-randomized iStent: Implantation of one iStent in conjunction with cataract surgery, patients not randomized to group

SUMMARY:
The purpose of this study is to assess the long-term safety of the Glaukos® iStent® Trabecular Micro-Bypass Stent Model GTS100R/L in subjects previously enrolled in Glaukos Study GC-003.

DETAILED DESCRIPTION:
The goal of this study was to demonstrate that use of this device in conjunction with cataract surgery did not result in a rate of sight-threatening adverse events, after 5 years of implantation that was higher than the rate of sight-threatening adverse events that occurred after cataract surgery alone, by more than a non-inferiority margin of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Subjects previously enrolled in Glaukos Study GC-003 who are able and willing to participate in this extended follow-up study

Exclusion Criteria:

* Subjects previously enrolled in Glaukos Study GC-003 who are not able or willing to participate in this extended follow-up study
* Patients not previously enrolled in Glaukos Study GC-003

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extended follow-up of subjects previously enrolled in Glaukos Study GC-003
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Wells, PharmD, MBA, Study Director — Glaukos Corporation; Jay Katz, MD, Study Chair — Wills Eye Institute; Thomas Jefferson University
Locations (26):
- United States (26):
  - Beverly Hills, California
  - Petaluma, California
  - Sacramento, California
  - San Clemente, California
  - Santa Maria, California
  - Parker, Colorado
  - Boynton Beach, Florida
  - Miami, Florida
  - Tampa, Florida
  - Morrow, Georgia
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Saint Joseph, Michigan
  - Bloomington, Minnesota
  - Edina, Minnesota
  - Independence, Missouri
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Brookville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Beaumont, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Randomized iStent | Randomized Cataract Surgery | Non-randomized iStent
Started | 51 | 35 | 22
Completed | 51 | 35 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Note: 108 of the subjects in the original pivotal trial participated in the follow-up study. There were 51 subjects from the randomized stent group, 35 from the cataract only group, and 22 from the non-randomized stent group who participated in this study
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized iStent | Randomized Cataract Surgery | Non-randomized iStent | Total
Number analyzed (Participants) | 51 | 35 | 22 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (7.7) | 69 (8.4) | 71 (8.6) | 71 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 10 | 57
  Male | 26 | 13 | 12 | 51
Region of Enrollment [Number; unit: participants]
  United States | 51 | 35 | 22 | 108

OUTCOME MEASURES:

1. Primary Outcome: Rate of Sight-threatening Adverse Events
Description: The primary endpoint is the occurrence of sight-threatening adverse events. The rate of sight-threatening adverse events at each visit will be calculated for the three treatment groups (randomized control group, randomized iStent group, and non-randomized iStent group) separately. The summary will also be performed for pooling the randomized iStent and non-randomized iStent group.
Time Frame: 80 Month average
Measure: Number; unit: percentage of subjects
Arm/Group | Randomized iStent | Randomized Cataract Surgery | Non-randomized iStent
Number analyzed (Participants) | 51 | 35 | 22
percentage of subjects | 27.8 | 45.7 | 34.3

ADVERSE EVENTS:
Arm/Group | Randomized iStent | Randomized Cataract Surgery | Non-randomized iStent
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/122 | 0/46
Other Adverse Events (participants affected / at risk) | 13/111 | 15/122 | 6/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized iStent (N=111) | Randomized Cataract Surgery (N=122) | Non-randomized iStent (N=46)
Age-related macular degeneration or worsening of AMD (Eye disorders) | 7 (8) | 6 (6) | 1 (1)
Epiretinal membrane (Eye disorders) | 4 (4) | 2 (4) | 5 (5)
Loss of BCVA greater or equal to 3 lines (Eye disorders) | 2 (2) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days